CLINICAL TRIAL: NCT05066659
Title: Relationship Between Balance Performance and Corticomotor Inhibition in Individuals With Parkinsons' Disease
Brief Title: Balance Performance and Corticomotor Inhibition in PD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM110122F
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Transcranial magnetic stimulation; Motor cortex; Corticomotor inhibition; Balance performance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postural instability is one of the motor features of Parkinson's disease (PD). Most patients will develop balance dysfunction, and they may get worse with disease progression. According to previous studies, people with PD had abnormal changes in corticomotor excitability, especially disinhibition in the primary motor cortex (M1). Some evidence had shown that the cortical function in the M1 is crucial for the pathophysiology of the underlying motor symptoms in PD. Furthermore, neurostimulation over the M1 could modulate the corticomotor excitability in individuals with PD, and then improve their motor and also balance performance. However, whether the impaired corticomotor inhibition relates to balance dysfunction in people with PD is still unknown. In this study, the purpose is to investigate the possible relationship between corticomotor inhibition and balance performance in individuals with PD. However, the postural position during TMS measurement may affect the corticomotor excitability. To further establish the above-mentioned relationship, the secondary purpose is to explore and confirm whether the postural position will influence the correlation.

ELIGIBILITY:
Inclusion Criteria:

* the Hoehn and Yahr stage between 1 and 3
* age 40 to 80 years
* a stable treatment of anti-PD medications

Exclusion Criteria:

* any contraindications of TMS
* any injury histories or disorders affecting balance
* any neurosurgery experience
* neurologic conditions other than PD
* the Mini-mental State Examination (MMSE) score < 24

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-08 (Estimated); Primary Completion 2022-09-08 (Estimated); Study Completion 2022-09-08 (Estimated)

PRIMARY OUTCOMES:
Intracortical inhibition | 20 minutes
  Short-interval intracortical inhibition assessed by transcranial magnetic stimulation
Corticospinal inhibition | 20 minutes
  Cortical silent period assessed by transcranial magnetic stimulation
Static balance | 3 minutes
  Sharpened Romberg test
Dynamic balance | 5 minutes
  Functional reach test
Functional balance | 15 minutes
  Mini-Balance Evaluation Systems Test

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided